CLINICAL TRIAL: NCT02562599
Title: Study Of Induction Chemotherapy Followed by Concurrent Chemoradiotherapy With Raltitrexed-Cisplatin for Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Chemoradiotherapy for Patients With Locally Advanced Nasopharyngeal Carcinoma Using Raltitrexed-Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HU DESHENG, Associate dean, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Radiotherapy center-001
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Induction Chemotherapy; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — raltitrexed; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- drug:raltitrexed safety and efficacy (Experimental): To receive the safety and efficacy of raltitrexed-cisplatin neoadjuvant chemotherapy followed by concurrent chemoradiotherapy with raltitrexed-cisplatin
  Interventions:
  Neochemotherapy (Induction Chemotherapy) Drugs: raltitrexed-cisplatin (Raltitrexed, 2.5mg/m2, IV in 15 minutes, d1; Cisplatin, 25mg/m2, IV, d1-3.Cycled every 21 days for 2 cycles).
  Concurrent Chemotherapy Drugs: raltitrexed-cisplatin (Raltitrexed, 2.5mg/m2, IV in 15 minutes, d1; Cisplatin, 25mg/m2, IV, d1-3.Cycled every 21 days for 2 cycles) .
  Radiation: Intensity-modulated radiotherapy (IMRT)
  Interventions: Drug: raltitrexed-cisplatin; Radiation: Intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: raltitrexed-cisplatin — Patients receive raltitrexed-cisplatin neoadjuvant chemotherapy every three weeks for two cycles, then receive raltitrexed -cisplatin concurrent chemoradiotherapy every three weeks for two cycles
  Other Names: Tomudex
Radiation: Intensity-modulated radiotherapy (IMRT) — Patients receive raltitrexed -cisplatin concurrent chemoradiotherapy every three weeks for two cycles

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of raltitrexed and cisplatin neoadjuvant chemotherapy followed by concurrent radiotherapy with raltitrexed and cisplatin in patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Although concurrent chemoradiation is the standard treatment modality for locally advanced nasopharyngeal carcinoma (NPC), high incidences of distant metastases and severe treatment related toxicities have become an obstacle to be overcome. A phase Ⅱ study conducted by Hui et al. showed that neoadjuvant chemotherapy followed by concurrent chemoradiotherapy was superior to the standard concomitant chemoradiation in terms of the 3-year OS without significantly exacerbating the acute toxicities.

At present, PF regimen has been considered as the most classic chemotherapy regimen of nasopharyngeal carcinoma (NPC), but its efficiency is about 40%-60% , and always with severe gastrointestinal reactions, renal toxicity and oral mucosa reaction. Therefore, it is imperative to find a more safe and effective chemotherapy regimen.

Raltitrexed is a specific thymidylate synthase inhibitor with a convenient administration schedule,acceptable and manageable toxicity, radiosensitising properties. It may offer advantages compared with standard 5-FU chemotherapy regimens used in locally advanced NPC.

Therefore, the investigators initiated this study to evaluate the efficacy and safety of raltitrexed and cisplatin neoadjuvant chemotherapy followed by concurrent radiotherapy with raltitrexed and cisplatin in patients with locally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed nasopharyngeal carcinoma, including WHO III
2. Newly diagnosed T3-4 or any TN2-3 locally advanced nasopharyngeal carcinoma
3. At least one measurable lesion (according to the RECIST1.1)
4. female and male,18-70 years of age
5. ECOG performance status of 0-1
6. Life expectancy of more than 3 months
7. Without radiotherapy or chemotherapy
8. Adequate organ function including the following:

   Platelets count >= 100 * 109/l Absolute neutrophil count (ANC) >= 2.0 * 109/l Hemoglobin >= 90 g/l Total bilirubin <= 1.5ULN AST and ALT <= 2.5ULN,if there is liver metastasis , AST and ALT <= 5ULN Serum creatine <= 1.5ULN
9. Signed and dated informed consent.

Exclusion Criteria:

1. Before or at the same time any second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
2. Evidence of distant metastasis
3. Taboos of chemotherapy or radiotherapy(such as heart failure, angina pectoris, or cardiac arrhythmia.et al) Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
4. Pregnant or breast-feeding females
5. Abuse of psychiatric drugs or dysphrenia
6. Prior chemotherapy with raltitrexed or cisplatin
7. Allergic to clinical drugs
8. Participation in clinical trials for other anti-tumor drugs in 4 weeks
9. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | up to 12 weeks

SECONDARY OUTCOMES:
OS(Overall Survival) | 2 years
TTP（Time To Progression） | 2 years
DCR (Disease Control Rate) | 6 weeks after induction chemotherapy; 4 weeks and 12 weeks after radiotherapy.
QOL（Quality Of Life） | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Desheng Hu, M.D., Principal Investigator — Associate dean
Locations (1):
- Hubei Cancer hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
There are not enough people participated in the treatment.